CLINICAL TRIAL: NCT01251900
Title: BRCA1 and BRCA2 Mutations and Triple Negative Disease in Hispanic/Latino Breast Cancer Subjects
Brief Title: BRCA Mutations in Latinas
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911035; 11-C-N035
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-09-25

CONDITIONS: Breast Neoplasms
Keywords: Triple Negative Disease; BRCA1; BRCA2; Hispanic/Latino; Breast Cancer; Natural History
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Hispanic women, over the age of 18, with breast cancer will be eligible.

SUMMARY:
Background:

- BRCA1 and BRCA2 gene mutations have been linked to a higher risk of developing breast cancer and other cancers, and may be associated with types of breast cancer that are more difficult to treat and more likely to recur. New cancer treatments are being developed specifically to treat individuals who have these gene mutations. However, more information is needed about the prevalence of these mutations in minority populations, including Hispanic/Latino populations. To study these populations, researchers are interested in collecting genetic material (DNA) and medical history information from Hispanic/Latino women who have been diagnosed with breast cancer.

Objectives:

- To collect saliva samples and medical and family history information from Hispanic/Latino women with breast cancer.

Eligibility:

- Hispanic/Latino women at least 18 years of age who have been diagnosed with breast cancer.

Design:

* Participants will complete a questionnaire with information about place of birth, languages spoken by parents and grandparents, and information about their breast cancer diagnosis.
* Participants will provide a saliva sample (2 to 3 tablespoons) for analysis.
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
BACKGROUND:

* Mutations in the BRCA1 and BRCA2 genes predispose to breast and ovarian cancer, and are increasingly recognized in prostate and pancreatic cancers.
* Basal/ Triple negative breast cancer is associated with BRCA mutations in some ethnicities.However the link between BRCA gene mutations and Basil/ triple negative disease in Hispanic/ Latino women is not known.
* Common recurrent mutations in BRCA1 and BRCA2 exist in Hispanic/ Latino communities.
* New therapies such as PARP inhibitors may be particularly effective in BRCA mutation carriers.
* Therefore a unique opportunity exists to identify women in this underserved minority that may be eligible for and benefit from new targeted therapies.

OBJECTIVES:

- The primary objective is to collect saliva samples and histology data from up to 2000 Hispanic/ Latino subjects with breast cancer as a source of DNA, and to analyze the BRCA1 and BRCA2 genes..

ELIGIBILITY:

- All Hispanics females, over the age of 18, with breast cancer will be eligible.

DESIGN:

- Natural history study of 2000 Hispanic/Latino women with breast cancer, 1000 with triple

negative disease, 1000 without.

* Obtain clinical pathology reports and relevant history data on all subjects.
* Analyze recurrent BRCA1 and BRCA2 mutations

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patient must be self-identified of Hispanic/Latino origin.
* Patients must have histologically or cytologically confirmed diagnosis of breast cancer.
* Age greater than or equal to 18 years.
* Ability to understand and the willingness to sign a written informed consent document.
* Must be willing and able to provide a saliva sample, answer questionnaire data online or complete a paper questionnaire, and request a copy of their pathology report.

EXCLUSION CRITERIA:

- Males and subjects under the age of 18.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2011-07-07 (Actual)

PRIMARY OUTCOMES:
Collection of saliva from 2000 probands | Every six months

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Dean, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Southwest Cancer Center, Lubbock; Texas Tech University, Lubbock, Texas, United States

REFERENCES:
- [Background] Dean M, Boland J, Yeager M, Im KM, Garland L, Rodriguez-Herrera M, Perez M, Mitchell J, Roberson D, Jones K, Lee HJ, Eggebeen R, Sawitzke J, Bass S, Zhang X, Robles V, Hollis C, Barajas C, Rath E, Arentz C, Figueroa JA, Nguyen DD, Nahleh Z. Addressing health disparities in Hispanic breast cancer: accurate and inexpensive sequencing of BRCA1 and BRCA2. Gigascience. 2015 Nov 4;4:50. doi: 10.1186/s13742-015-0088-z. eCollection 2015. PMID 26543556